CLINICAL TRIAL: NCT03318432
Title: Stroke Recovery Initiative - Stroke Registry
Brief Title: Stroke Recovery Initiative - Registry for Stroke Research Studies
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 11-07808
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Acute Stroke; Ischemic Stroke; Hemorrhagic Stroke; Subarachnoid Hemorrhage; Cerebral Ischemia; Cerebral Infarction; Cerebral Stroke; Cerebral Vascular Accident
Keywords: Stroke; Acute Stroke; Ischemic Stroke; Hemorrhagic Stroke; Cerebral Ischemia; Cerebral Infarction; Cerebral Stroke; Cerebral Vascular Accident; Stroke Recovery
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Subarachnoid Hemorrhage; Brain Ischemia; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Stroke Recovery Initiative is a nation-wide participant recruitment registry that connects people who have had a stroke with researchers who are working to develop new approaches to improve recovery after stroke.

DETAILED DESCRIPTION:
The Stroke Recovery Initiative at UCSF is designed to help people who have had a stroke to connect with researchers who are applying the latest science and technology to develop new treatments for stroke recovery. Anyone who is 18 years of age or older and has had a stroke may submit a survey to join. The self-reported information on the survey will be used to match participants to current or future stroke research studies and study personnel for each specific study may contact participants for further screening. Some studies are recruiting participants nationally, not just in the San Francisco Bay Area.

ELIGIBILITY:
* 18 years of age or older
* Have suffered a stroke
* Have ongoing symptoms as a result of the stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2013-02-09 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Total Enrollment | 5 years
  Total Number of Participants in the Registry

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S. Kim, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stroke Recovery Initiative — https://strokerecoveryinitiative.ucsf.edu/